CLINICAL TRIAL: NCT00665912
Title: Platelet-Rich and Concentrated Platelet Poor Plasma to Reduce Air Leak Post Lobectomy: A Randomized Controlled Trial
Brief Title: Platelet-Rich and Concentrated Platelet-Poor Plasma to Reduce Air Leak Post-Lobectomy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBI-004
Record Dates: First submitted 2008-04-21; First posted 2008-04-24 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Standard post-lobectomy wound care plus use of PRP and PPPc in the thoracic cavity.
  Interventions: Procedure: Standard post-lobectomy wound care plus use of PRP and PPPc prepared by GPS and Plasmax respectively
- 2 (Active Comparator): Standard post-lobectomy wound care in the thoracic cavity
  Interventions: Procedure: Standard post-lobectomy wound care

INTERVENTIONS:
Procedure: Standard post-lobectomy wound care plus use of PRP and PPPc prepared by GPS and Plasmax respectively — GPS is used to create the platelet rich plasma (PRP). Plasmax is used to create the concentrated platelet-poor plasma (PPPc). Both PRP and PPPc will be used for wound care in the thoracic cavity post-lobectomy.
  Arms: 1
Procedure: Standard post-lobectomy wound care — Standard post-lobectomy wound care
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the use of platelet-rich plasma (PRP) and concentrated platelet-poor plasma (PPPc) can reduce the duration of post-operative air leak after lobectomy for lung tumours.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a lobectomy

Exclusion Criteria:

* Pneumonectomy
* Sleeve lobectomy
* Determination of unresectability (prior to the initiation of lobectomy)
* Wedge resection alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative air leak | Every 4 hours of postop hospital stay, between 4-6 weeks postop

SECONDARY OUTCOMES:
Incidence of air leak, Prolonged air leak (> days), Complications | Every 4 hours of postop hospital stay, between 4-6 weeks postop

CONTACTS AND LOCATIONS:
Overall Officials: Richard Inculet, MD, FRCSC, FACS, Principal Investigator — Western University, Canada; Darrin Payne, MD, Study Chair — Western University, Canada; Dalilah Fortin, MD, Study Chair — Western University, Canada; Richard Malthaner, MD, Study Chair — Western University, Canada; Robert Humphrey, MD, Study Chair — Western University, Canada
Locations (1):
- University of Western Ontario: Division of Thoracic Surgery, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No